CLINICAL TRIAL: NCT01987453
Title: An Open-Label, Multicenter Study To Evaluate The Efficacy And Safety Of Sofosbuvir/Ledipasvir Fixed-Dose Combination ± Ribavirin For 12 or 24 Weeks In Chronic Genotype 1 HCV Infected Subjects Who Participated In A Prior Gilead-Sponsored HCV Treatment Study
Brief Title: Ledipasvir/Sofosbuvir Fixed-Dose Combination ± Ribavirin in Participants With Chronic Genotype 1 HCV Who Participated in a Prior Gilead-Sponsored HCV Treatment Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1118; 2014-001245-24 (EudraCT Number)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2016-11

CONDITIONS: HCV Infection
Keywords: genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LDV/SOF+RBV 12 weeks (Group 1) (Experimental): Participants who failed a prior SOF+RBV ± pegylated interferon (Peg-IFN) regimen will receive LDV/SOF FDC plus RBV for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF 24 weeks (Group 2) (Experimental): Participants who failed a prior LDV/SOF ± RBV regimen will receive LDV/SOF FDC for 24 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 24 weeks (Group 3) (Experimental): Participants with advanced compensated or decompensated cirrhosis who failed a prior SOF+RBV regimen will receive LDV/SOF FDC plus RBV for 24 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — Tablet(s) administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — Tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Participants in the LDV/SOF+RBV 24 weeks group will dose adjust RBV according to hemoglobin and renal status as stated in the RBV package insert.
  Arms: LDV/SOF+RBV 12 weeks (Group 1); LDV/SOF+RBV 24 weeks (Group 3)

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) with or without ribavirin (RBV) in participants with chronic genotype 1 hepatitis C virus (HCV) infection who have participated in a prior Gilead-sponsored HCV treatment study, and who did not achieve sustained virologic response (SVR24), defined as HCV RNA < lower limit of quantification (LLOQ) 24 weeks after last dose of study drug (SVR24).

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* Infection with HCV genotype 1
* HCV RNA > LLOQ at screening
* Participation in a prior Gilead-sponsored study
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male
* Must be of generally good health, with the exception of chronic HCV infection, as determined by the Investigator
* Must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments

Key Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Co-infection with HIV or hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation (Groups 1 and 2 only)
* Hepatocellular carcinoma (HCC)
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (41):
- United States (37):
  - Beverly Hills, California
  - La Jolla, California
  - Los Angeles, California
  - Oceanside, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Downers Grove, Illinois
  - Indianapolis, Indiana
  - Bowling Green, Kentucky
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Hillsborough, New Jersey
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Manhasset, New York
  - New York, New York
  - Asheville, North Carolina
  - Winston-Salem, North Carolina
  - Philadelphia, Pennsylvania
  - Germantown, Tennessee
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Camperdown, New South Wales, Australia
- Clichy, France
- San Juan, Puerto Rico
- Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Background] Lawitz E, Pockros PJ, Yang JC, Pang PS, Zhu Y, Svarovskaia E, et al. Ledipasvir/sofosbuvir regimens for the retreatment of patients who failed sofosbuvir-based regimens [Abstract 10868]. Presented at: The 25th Conference of the Asian Pacific Association for the Study of Liver (APASL); 2016 February 20-24; Tokyo, Japan.
- [Background] Lawitz E, Flamm S, Yang JC, Pang PS, Zhu Y, Svarovskaia E, et al. Retreatment of patients who failed 8 or 12 weeks of ledipasvir/sofosbuvir-based regimens with ledipasvir/sofosbuvir for 24 weeks [Abstract 1627]. Presented at: The 50th Annual Congress of the European Association for the Study of Liver: The International Liver Congress (EASL); 2015 April 22-26; Vienna, Austria
- [Result] Wyles D, Pockros P, Morelli G, Younes Z, Svarovskaia E, Yang JC, Pang PS, Zhu Y, McHutchison JG, Flamm S, Lawitz E. Ledipasvir-sofosbuvir plus ribavirin for patients with genotype 1 hepatitis C virus previously treated in clinical trials of sofosbuvir regimens. Hepatology. 2015 Jun;61(6):1793-7. doi: 10.1002/hep.27814. Epub 2015 Apr 27. PMID 25846014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the US, Australia, and Spain. The first participant was screened on 30 July 2014. The last study visit occurred on 12 November 2015.
Pre-assignment Details: 101 participants were screened.
Groups:
- LDV/SOF + RBV 12 Weeks (Group 1): Participants who failed a prior sofosbuvir (SOF) + ribavirin (RBV) ± pegylated interferon (Peg-IFN) regimen received ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet administered orally once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- LDV/SOF 24 Weeks (Group 2): Participants who failed a prior LDV/SOF±RBV regimen received LDV/SOF FDC (90/400 mg) tablet administered orally once daily for 24 weeks
- LDV/SOF + RBV 24 Weeks (Group 3): Participants with advanced compensated or decompensated cirrhosis who failed a prior SOF+RBV regimen received LDV/SOF FDC (90/400 mg) tablet administered orally once daily + RBV (adjusted for hemoglobin and renal status) for 24 weeks
Period: Overall Study
Arm/Group | LDV/SOF + RBV 12 Weeks (Group 1) | LDV/SOF 24 Weeks (Group 2) | LDV/SOF + RBV 24 Weeks (Group 3)
Started | 51 | 41 | 8
Completed | 50 | 29 | 7
Not Completed | 1 | 12 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 12 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Groups:
- LDV/SOF + RBV 12 Weeks (Group 1): Participants who failed a prior SOF+RBV ± Peg-IFN regimen received ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet administered orally once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF + RBV 12 Weeks (Group 1) | LDV/SOF 24 Weeks (Group 2) | LDV/SOF + RBV 24 Weeks (Group 3) | Total
Number analyzed (Participants) | 51 | 41 | 8 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (8.7) | 58 (6.9) | 61 (6.7) | 57 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 7 | 1 | 28
  Male | 31 | 34 | 7 | 72
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 8 | 10 | 1 | 19
  White | 43 | 31 | 7 | 81
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 4 | 5 | 0 | 9
  Not Hispanic or Latino | 47 | 36 | 8 | 91
Region of Enrollment [Number; unit: participants]
  United States | 51 | 41 | 4 | 96
  Australia | 0 | 0 | 1 | 1
  Spain | 0 | 0 | 3 | 3
Prior HCV Treatment Experience [Number; unit: Particiapants]
  SOF+PEG+RBV | 25 | 0 | 0 | 25
  SOF+RBV | 20 | 0 | 8 | 28
  LDV/SOF | 0 | 18 | 0 | 18
  LDV/SOF+RBV | 0 | 15 | 0 | 15
  LDV/SOF+GS-9669 | 0 | 8 | 0 | 8
  Without SOF | 6 | 0 | 0 | 6
IL28B [Number; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 4 | 3 | 0 | 7
    CT | 33 | 27 | 7 | 67
    TT | 14 | 11 | 1 | 26
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.58) | 6.2 (0.62) | 5.6 (0.44) | 6.2 (0.61)
HCV RNA Category [Number; unit: Participants]
  < 800,000 IU/mL | 13 | 11 | 6 | 30
  >= 800,000 IU/mL | 38 | 30 | 2 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study treatment.
Time Frame: Post-treatment Week 12
Population: Full Analysis Set: participants enrolled into the study and received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Groups:
- LDV/SOF + RBV 12 Weeks (Group 1): Participants who failed a prior SOF+RBV ± Peg-IFN regimen received LDV/SOF (90/400 mg) FDC tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- LDV/SOF 24 Weeks (Group 2): Participants who failed a prior LDV/SOF ± RBV regimen received LDV/SOF FDC (90/400 mg) tablet administered orally once daily for 24 weeks
Arm/Group | LDV/SOF + RBV 12 Weeks (Group 1) | LDV/SOF 24 Weeks (Group 2) | LDV/SOF + RBV 24 Weeks (Group 3)
Number analyzed (Participants) | 51 | 41 | 8
Percentage of participants | 98.0 | 70.7 | 100.0

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 Weeks
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Groups:
- LDV/SOF 24 Weeks (Group 2): Participants who failed a prior LDV/SOF± RBV regimen received LDV/SOF FDC (90/400 mg) tablet administered orally once daily for 24 weeks
- LDV/SOF + RBV 24 Weeks (Group 3): Participants with advanced compensated or decompensated cirrhosis who failed a prior SOF + RBV regimen received LDV/SOF FDC (90/400 mg) tablet administered orally once daily + RBV (adjusted for hemoglobin and renal status) for 24 weeks
Arm/Group | LDV/SOF + RBV 12 Weeks (Group 1) | LDV/SOF 24 Weeks (Group 2) | LDV/SOF + RBV 24 Weeks (Group 3)
Number analyzed (Participants) | 51 | 41 | 8
Percentage of participants | 5.9 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | LDV/SOF + RBV 12 Weeks (Group 1) | LDV/SOF 24 Weeks (Group 2) | LDV/SOF + RBV 24 Weeks (Group 3)
Number analyzed (Participants) | 51 | 41 | 8
Percentage of participants
  SVR4 | 98.0 | 73.2 | 100.0
  SVR24 | 98.0 | 70.7 | 100.0

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ While on Treatment
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | LDV/SOF + RBV 12 Weeks (Group 1) | LDV/SOF 24 Weeks (Group 2) | LDV/SOF + RBV 24 Weeks (Group 3)
Number analyzed (Participants) | 51 | 41 | 8
Percentage of participants
  Week 1 | 23.5 | 31.7 | 0
  Week 4 | 98.0 | 95.1 | 100.0
  Week 8 | 100.0 | 100.0 | 100.0
  Week 12 | 100.0 | 100.0 | 100.0
  Week 16 | NA — Treatment for this group was 12 weeks only. | 97.6 | 100.0
  Week 20 | NA — Treatment for this group was 12 weeks only. | 97.6 | 100.0
  Week 24 | NA — Treatment for this group was 12 weeks only. | 100.0 | 100.0

5. Secondary Outcome: Change in HCV RNA From Baseline
Time Frame: Baseline to Week 8
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF + RBV 12 Weeks (Group 1) | LDV/SOF 24 Weeks (Group 2) | LDV/SOF + RBV 24 Weeks (Group 3)
Number analyzed (Participants) | 51 | 41 | 8
log10 IU/mL
  Week 1 | -4.47 (0.500) | -4.40 (0.535) | -3.75 (0.878)
  Week 4 | -5.07 (0.565) | -5.06 (0.600) | -4.47 (0.441)
  Week 8 | -5.09 (0.583) | -5.08 (0.617) | -4.47 (0.441)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit confirmed with 2 consecutive values or last available posttreatment measurement
Time Frame: Up to posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | LDV/SOF + RBV 12 Weeks (Group 1) | LDV/SOF 24 Weeks (Group 2) | LDV/SOF + RBV 24 Weeks (Group 3)
Number analyzed (Participants) | 51 | 41 | 8
Percentage of participants
  On treatment Virologic Failure | 0 | 2.4 | 0
  Relapse | 2.0 | 27.5 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Groups:
- LDV/SOF + RBV 12 Weeks (Group 1): Participants who failed a prior SOF+RBV ± Peg-IFN regimen received LDV/SOF (90/400 mg) FDC tablet administered orally once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- LDV/SOF 24 Week (Group 2): Participants who failed a prior LDV/SOF±RBV regimen received LDV/SOF FDC (90/400 mg) tablet administered orally once daily for 24 weeks
- LDV/SOF + RBV 24 Week (Group 3): Participants with advanced compensated or decompensated cirrhosis who failed a prior SOF+RBV regimen received LDV/SOF FDC (90/400 mg) tablet administered orally once daily + RBV (adjusted for hemoglobin and renal status) for 24 weeks
Arm/Group | LDV/SOF + RBV 12 Weeks (Group 1) | LDV/SOF 24 Week (Group 2) | LDV/SOF + RBV 24 Week (Group 3)
Serious Adverse Events (participants affected / at risk) | 2/51 | 2/41 | 2/8
Other Adverse Events (participants affected / at risk) | 37/51 | 16/41 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF + RBV 12 Weeks (Group 1) (N=51) | LDV/SOF 24 Week (Group 2) (N=41) | LDV/SOF + RBV 24 Week (Group 3) (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF + RBV 12 Weeks (Group 1) (N=51) | LDV/SOF 24 Week (Group 2) (N=41) | LDV/SOF + RBV 24 Week (Group 3) (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Fatigue (General disorders) | 13 | 4 | 3
Oedema (General disorders) | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 2
Anal abscess (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 3 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 11 | 6 | 0
Depression (Psychiatric disorders) | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 3 | 2
Irritability (Psychiatric disorders) | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years